CLINICAL TRIAL: NCT06439563
Title: A Multicenter, Parallel, Double-blind, Randomized, Active-controlled, Non-inferiority, Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of JP-1366 Treatment in the Prevention of (NSAIDs)-Induced Peptic Ulcers
Brief Title: Study to Evaluate the Efficacy and Safety of JP-1366 in the Prevention of NSAIDs-Induced Peptic Ulcers
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Onconic Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JP-1366-304
Record Dates: First submitted 2024-05-22; First posted 2024-06-03 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Peptic Ulcer
MeSH Terms: conditions — Peptic Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JP-1366 10 mg (Experimental)
  Interventions: Drug: JP-1366 10 mg; Drug: Lanston Capsule 15 mg placebo
- Lanston Capsule 15 mg (Active Comparator)
  Interventions: Drug: Lanston Capsule 15 mg; Drug: JP-1366 10 mg placebo

INTERVENTIONS:
Drug: JP-1366 10 mg — JP-1366 10 mg, tablet, orally once a day for up to 24 weeks
  Arms: JP-1366 10 mg
Drug: Lanston Capsule 15 mg — Lanston Capsule 15 mg orally once a day for up to 24 weeks
  Arms: Lanston Capsule 15 mg
Drug: JP-1366 10 mg placebo — JP-1366 10 mg placebo, tablet, orally once a day for up to 24 weeks
  Arms: Lanston Capsule 15 mg
Drug: Lanston Capsule 15 mg placebo — Lanston Capsule 15 mg placebo, orally once a day for up to 24 weeks
  Arms: JP-1366 10 mg

SUMMARY:
The sutdy aims to to demonstrate the non-inferiority of JP-1366 10 mg compared to Lanston Capsule 15 mg in preventing NSAIDs-induced peptic ulcers and to compare/evaluate the efficacy and safety of JP-1366 10 mg.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male/female aged 19 years or older as of the date of obtaining consent
2. Those who are diagnosed with musculoskeletal diseases such as rheumatoid arthritis, osteoarthritis, ankylosing spondylitis, or other diseases at the time of screening and require continuous administration of NSAIDs for 24 weeks or more
3. Those with one or more of the following risk factors for ulcer development at the time of screening
4. Subjects who fully understand this study and voluntarily signed the informed consent form.

Exclusion Criteria:

1. Those who cannot undergo upper gastrointestinal endoscopy
2. At the time of screening, those who were confirmed to have active stage ulcers (A1, A2) or healing stage ulcers (H1, H2) in the stomach or duodenum according to the Sakita-Miwa Classification*
3. Those with a confirmed history of malignant tumor within 5 years
4. Those with a confirmed history of signal symptoms suggestive of malignant disease of the gastrointestinal tract
5. Those who need to continuously take corticosteroids, antiplatelet agents, and anticoagulants during this study (however, the following cases are permitted):
6. Pregnant and lactating women or those with a positive pregnancy test result at screening
7. Those who participated in another study and were administered investigational products or had medical devices applied at least once within 4 weeks from the screening visit(Visit 0)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative proportion of subjects who developed peptic ulcers | at 24 weeks after administration of investigational products

SECONDARY OUTCOMES:
Proportion of subjects with gastric or duodenal endoscopic bleeding | at 24 weeks after administration of investigational products

CONTACTS AND LOCATIONS:
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No